CLINICAL TRIAL: NCT01452048
Title: Relationship Between Systemic Fatty Acid Availability and Insulin Sensitivity
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Associate Professor, Movement Science, School of Kinesiology, University of Michigan
Other Study IDs: R01 DK077966 - OC; R01DK077966 (NIH)
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Obesity
Keywords: insulin sensitivity; fatty acid metabolism
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — frozen tissue, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obese Sedentary Adults, but otherwise healthy

SUMMARY:
The investigators specific aim is to compare the relationship between systemic fatty acid availability and insulin sensitivity in a relatively homogenous population of obese adults. The investigators anticipate 1) greater systemic fatty acid availability will be associated with lower insulin sensitivity and 2) greater systemic fatty acid availability will be associated with greater accumulation of fatty acid intermediates and pro-inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index [BMI]: 35-45 kg/m2; All women must be pre-menopausal; Non-exerciser (no regularly planned exercise/physical activity)

Exclusion Criteria:

* Weight instability ≥ ±5 lbs. in past month; medications known to affect lipid and/or glucose metabolism; Pregnancy or actively breast feeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: UM Health System patients from Dr. Amy Rothberg and colleagues UM Investigational Weight Management Clinic (IWMC) Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2011-09; Primary Completion 2016-05-26 (Actual); Study Completion 2016-05-26 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | 2-3 hours
  A hyperinsulinemic-euglycemic clamp will be used to assess peripheral insulin sensitivity

SECONDARY OUTCOMES:
Resting Metabolic Rate | 20-30 min

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Horowitz, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- Michigan Clincal Research Unit, Ann Arbor, Michigan, United States